CLINICAL TRIAL: NCT00449683
Title: Antidepressant Induced Excessive Sweating: Measurement and Treatment With Terazosin
Brief Title: Excessive Sweating Caused by Antidepressants: Measurement and Treatment With Terazosin
Acronym: ADIES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06F.275
Record Dates: First submitted 2007-03-19; First posted 2007-03-20 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Hyperhidrosis
Keywords: Depressive Disorders; Excessive Sweating; Sweating caused by antidepressants for those a depressive disorder
MeSH Terms: conditions — Hyperhidrosis; Depressive Disorder | interventions — Terazosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- terazosin (Experimental): open-label treatment group
  Interventions: Drug: terazosin

INTERVENTIONS:
Drug: terazosin — off-label use of terazosin to treat antidepressant-induced sweating
  Other Names: Hytrin

SUMMARY:
The study consists of measurement of antidepressant-induced excessive sweating and its treatment with an experimental medication, terazosin (approved for hypertension), that will be added to the antidepressant. This study is for people who take an antidepressant due to a depressive disorder. This is an open-label study (no placebo group) that will last 5 weeks, with one week of baseline measurement and four weeks of treatment with the study medication. The study is based on the hypothesis that terazosin will be effective in reducing the severity of excessive sweating caused by antidepressant treatment, and will have minimal side-effects.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 75 years
2. Clinical diagnosis of a Depressive disorder (Diagnostic and Statistical Manual of Mental Disorders - IV-TR)
3. Presence of excessive sweating by self-report
4. The excessive sweating started after initiation of an antidepressant and, if treatment with the antidepressant was interrupted, did not persist for more than 4 weeks during that interruption
5. Treatment with the antidepressant is deemed to be clinically necessary due to substantial benefit from this antidepressant, and failure to respond to or tolerate an alternative
6. Excessive sweating has persisted for at least 4 weeks prior to baseline assessment
7. The excessive sweating is rated by the patient as at least moderately bothersome.
8. Episodes of excessive sweating occur at least twice a week for last 4 weeks

Exclusion Criteria:

1. Presence of another known disease that could potentially cause excessive sweating
2. Failure to respond to antiadrenergic (reducing activity of the sympathetic nervous system) treatment in the past
3. Blood pressure less than 110 mm Hg systolic at the screening or baseline visits
4. Orthostatic hypotension by history or on assessment at the screening or baseline visits (defined as a decrease of 10 mm Hg or greater after standing for 2 minutes).
5. Current antihypertensive treatment
6. History of significant cardiac disease, including coronary artery disease
7. Current use of phosphodiesterase type 5 inhibitors: sildenafil (ViagraTM), tadalafil (CialisTM), or vardenafil (LevitraTM)
8. History of priapism (persistent and painful erection)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
To study whether terazosin 1 to 4 mg/ day is effective in reducing antidepressant-induced sweating | 8 weeks
To test a novel device for ambulatory monitoring of sweating which is required to study this phenomenon since ADIES is usually episodic | 8 weeks

SECONDARY OUTCOMES:
To determine if the severity of sweating at baseline is correlated with baseline urinary norepinephrine levels | 8 weeks
To determine if response to treatment correlated with baseline urinary norepinephrine levels and with changes in these levels during the study. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rajnish Mago, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Department of Psychiatry, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mago R, Thase ME, Rovner BW. Antidepressant-induced excessive sweating: clinical features and treatment with terazosin. Ann Clin Psychiatry. 2013 Aug;25(3):186-92. Epub 2013 May 1. PMID 23638448